CLINICAL TRIAL: NCT03578978
Title: A Panel of Biomarkers in Diagnosing Late-onset Neonatal Sepsis and Necrotizing Enterocolitis in Sibu Hospital
Acronym: PISALONS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Sponsor
Other Study IDs: NMRR-17-2491-38373
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Neonatal SEPSIS; Necrotizing Enterocolitis
MeSH Terms: conditions — Neonatal Sepsis; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonates with suspected LONS and/or NEC: A group of 150 neonates with suspected LONS and/or NEC will be recruited. No intervention will be given to the subjects. Blood sampling will be obtained from subjects at 4 time points (Hour 0, 24, 48 and 72) for analysis of the sepsis biomarkers of interest.
  Interventions: Other: No intervention
- Healthy neonates: A group of 50 neonates who are clinically well, admitted to the NICU for reasons other than neonatal sepsis or NEC will be recruited into the study to explore the kinetics and concentrations of the panel of biomarkers in healthy subjects comparing to subjects with suspected LONS/NEC. No intervention will be given to the subjects. Blood sampling will be obtained from subjects at 4 time points (Hour 0, 24, 48 and 72) for analysis of the sepsis biomarkers of interest.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be given to study subjects. Only blood will be obtained from study subjects.

SUMMARY:
This is a cross-sectional study to evaluate the utilities of a panel of biomarkers (Procalcitonin, Interleukin-6, Serum Amyloid A and Apolipoprotein C2) versus the gold standard blood culture result diagnosing late-onset neonatal sepsis (LONS) and/or necrotizing enterocolitis (NEC). Neonates who meet the initial screening criteria for suspected LONS or NEC will be recruited into the study. A group of 50 neonates who are clinically well, admitted to the nursery or general ward for reasons other than neonatal sepsis or NEC will also be recruited into the study.

DETAILED DESCRIPTION:
The diagnosis of neonatal sepsis is challenging especially the very low birth weight infants as the signs and symptoms of sepsis are nonspecific and can be attributed to non-infected aetiologies including exacerbation of bronchopulmonary dysplasia, apnoea of prematurity and gastroesophageal reflux. Blood culture remains the gold standard for diagnosing septicaemia (either bacteremia or fungemia). However, its effectiveness in the population of preterm infants is compromised.Given the dire consequences of not treating the sepsis early, clinicians tend to have a low threshold for treatment. This leads to overuse of antimicrobials, promotion of antimicrobial resistance, exposure of infants to avoidable side effects from the antimicrobial treatment, prolonged hospitalisation and increased healthcare costs. Hence, there is a need for a clearly defined algorithm for diagnosing LONS and NEC. This study aims to examine the diagnostic utilities of a panel of sepsis biomarkers and explore if they can be incorporated into a diagnostic algorithm which hopefully, can be translated into clinical practice in the future.

ELIGIBILITY:
Neonates with suspected LONS/NEC

Inclusion Criteria:

* Infants with signs and symptoms suggestive of sepsis and/or NEC and requiring full sepsis screening and start of intravenous antibiotic(s), or a change of antibiotics (if already on)
* Infants with postnatal age greater than 72 hours and less than 28 days of life, of all gestation
* Parents of potential neonates who are willing to give written informed consent

Healthy subjects

Inclusion Criteria:

* Clinically well infants admitted to Sibu Hospital for reasons other than neonatal sepsis or NEC
* Infants with postnatal age greater than 72 hours and less than 28 days of life, of all gestation

Exclusion Criteria:

* Infants who have lethal or life-threatening congenital abnormalities
* Infants who have chromosomal abnormalities
* Infants who have hypoxic ischemic encephalopathy
* Infants who are on steroid treatment
* Infants who received blood transfusions
* Post-operative infants

Ages: 72 Hours to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates suspected of LONS and/or NEC admitted to the Neonatal Intensive Care Unit (NICU), Special Care Nursery (SCN) or Paediatric Medical 27 (PM27) wards in Sibu Hospital, Malaysia during the period of 1 July 2018 and 31 May 2020 will be screened for their eligibility. Apart from that, neonates admitted to Sibu Hospital for reasons other than neonatal sepsis or NEC will also be recruited into the study during the period of 1 June 2018 and 31 May 2020.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic utilities of biomarkers of interest in diagnosing LONS | Hour 0 to 72
  Diagnostic utilities of each individual biomarker (procalcitonin, interleukin-6, serum amyloid A and apolipoprotein C2) or in combination in diagnosing LONS
Diagnostic utilities of biomarkers of interest in diagnosing NEC | Hour 0 to 72
  Diagnostic utilities of each individual biomarker (procalcitonin, interleukin-6, serum amyloid A and apolipoprotein C2) or in combination in diagnosing LONS

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Hui Tan, Principal Investigator — Clinical Research Centre, Sarawak General Hospital, Malaysia
Locations (2):
- Malaysia (2):
  - Sarawak General Hospital, Kuching, Sarawak
  - Sibu Hospital, Sibu, Sarawak

IPD SHARING:
Plan to Share IPD: No